CLINICAL TRIAL: NCT07008352
Title: Examination of Preoperative and Postoperative Serum Amino Acid Metabolism in Individuals Undergoing Bariatric Surgery
Brief Title: Amino Acid Metabolism Before and After Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: Harran University (Other)
Responsible Party: Principal Investigator, Faik TATLI, Professor Dr, Harran University
Other Study IDs: Gerger
Record Dates: First submitted 2025-05-29; First posted 2025-06-06 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Obesity, Morbid
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples with DNA or without DNA will be retained
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Bariatric surgery patients (n=50): Participants in this group are adults (≥18 years old) with obesity who are scheduled to undergo bariatric surgery at Harran University Hospital. Blood samples will be collected at three time points: before surgery (baseline), and at 1 and 3 months postoperatively. Serum will be separated and stored at -80°C for subsequent amino acid profiling using LC-MS/MS.
  Interventions: Procedure: Blood sample collection for amino acid profiling
- Group 2: Healthy control participants (n=50): Participants in this group are healthy adults (≥18 years old) with no known history of obesity or chronic metabolic disease. A single blood sample will be collected at baseline. Serum samples will be analyzed using LC-MS/MS to determine amino acid profiles, which will be compared to those of the bariatric surgery group.
  Interventions: Procedure: Blood sample collection for amino acid profiling

INTERVENTIONS:
Procedure: Blood sample collection for amino acid profiling — Blood samples (5 mL) will be collected from participants in both groups. In the bariatric surgery group, samples will be collected at three time points: preoperatively, and at 1 and 3 months postoperatively. For the control group, a single sample will be obtained. Serum will be separated, stored at -80°C, and analyzed for free amino acid profiles using LC-MS/MS.

SUMMARY:
This observational study aims to investigate the changes in serum amino acid metabolism before and after bariatric surgery in obese individuals. Blood samples will be collected from 50 patients at baseline (preoperative), and at 1 and 3 months postoperatively. An additional 50 healthy individuals will serve as the control group. Amino acid profiling will be conducted using LC-MS/MS. The study seeks to determine how bariatric surgery affects metabolic pathways associated with amino acid regulation.

DETAILED DESCRIPTION:
Obesity is a major global health problem that significantly increases the risk of metabolic disorders. Bariatric surgery is one of the most effective interventions for sustained weight loss in morbidly obese patients. However, the metabolic effects of such surgery on amino acid profiles are not fully understood.

In this prospective observational study, a total of 100 participants will be enrolled: 50 patients undergoing bariatric surgery and 50 healthy controls. Serum samples will be collected from the patient group preoperatively, and at 1 and 3 months after surgery. The control group will provide one-time blood samples.

All serum samples will be centrifuged and stored at -80°C until analysis. Free amino acid profiles will be determined using liquid chromatography-tandem mass spectrometry (LC-MS/MS). The primary outcome is to assess the change in amino acid concentrations over time in surgical patients, and to compare them with healthy controls. Secondary analyses will explore correlations between amino acid levels and body mass index (BMI). Data analysis will be performed using SPSS and MetaboAnalyst 5.0.

This study will help clarify how bariatric surgery influences amino acid metabolism and may offer insights into the metabolic mechanisms underlying postoperative recovery and weight regulation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Diagnosed with obesity and scheduled for bariatric surgery (study group)
* Healthy individuals with normal BMI (control group)

Exclusion Criteria:

* Age <18 years
* History of metabolic or chronic systemic disease
* Pregnancy or lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will include 50 patients diagnosed with obesity and undergoing bariatric surgery, and 50 healthy adults with normal BMI values. All participants will be recruited from Harran University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2025-06-11 (Actual); Primary Completion 2025-10-02 (Actual); Study Completion 2025-11-03 (Actual)

PRIMARY OUTCOMES:
Change in serum free amino acid levels after bariatric surgery | Preoperative (baseline), 1 month postoperative, 3 months postoperative
  Amino acid concentrations will be measured in serum samples collected from bariatric surgery patients at baseline, 1 month, and 3 months postoperatively using LC-MS/MS. The outcome will assess time-dependent changes in the amino acid profile within the same individuals.

SECONDARY OUTCOMES:
Correlation between serum amino acid levels and body mass index (BMI) | Preoperative (baseline), 1 month postoperative, 3 months postoperative
  This outcome will evaluate the relationship between changes in serum amino acid concentrations and BMI values measured at baseline, 1 month, and 3 months after bariatric surgery. Pearson or Spearman correlation analyses will be performed.

CONTACTS AND LOCATIONS:
Locations (1):
- Veli Fahri Pehlivan, Sanliurfa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No